CLINICAL TRIAL: NCT06511180
Title: Introduction of Dispersible 3HP Formulations for TB Preventive Treatment in Children: a Multi-country Evaluation
Status: Not yet recruiting | Type: Observational
Sponsor: The Aurum Institute NPC (Other)
Collaborators: Johns Hopkins University (Other); KNCV Tuberculosis Foundation (Other); Clinton Health Access Initiative Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: AUR2-7-428; ERC.0004119 (Other: World Health Organisation)
Record Dates: First submitted 2024-07-16; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: TB - Tuberculosis; Household Contact; HIV; Children, Only
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Children <12 years who are eligible for TPT - HHC: No intervention. Clinic record review: Data will be retrospectively abstracted from routine medical files using a standardised data collection tool that will document TPT uptake and outcomes
- Policy makers/Program managers: No intervention. Qualitative study: We will recruit a purposive sample of policy makers, healthcare workers and caregivers who will be interviewed to evaluate buy-in and explore their insights and experiences on the different TPT regimens and formulations.
- Healthcare Workers: No intervention. Qualitative study: We will recruit a purposive sample of policy makers, healthcare workers and caregivers who will be interviewed to evaluate buy-in and explore their insights and experiences on the different TPT regimens and formulations.
- Caregivers: No intervention. Qualitative study: We will recruit a purposive sample of policy makers, healthcare workers and caregivers who will be interviewed to evaluate buy-in and explore their insights and experiences on the different TPT regimens and formulations.
- Pharmacy managers/pharmacists: No intervention. Clinic assessment: We will assess provider barriers and facilitators to prescribing the new dispersible 3HP (single dispersible formulations of isoniazid and rifapentine) through a survey tool which will collect information on the flow of TPT from national supply to the clinic and dispensing to the child.
- Procurement managers/Supply managers: No intervention. Clinic assessment: We will assess provider barriers and facilitators to prescribing the new dispersible 3HP (single dispersible formulations of isoniazid and rifapentine) through a survey tool which will collect information on the flow of TPT from national supply to the clinic and dispensing to the child.

SUMMARY:
The WHO has recommended TB preventive therapy (TPT) for children living with HIV (CLHIV) and household contacts of people living with TB, however, the scale-up and implementation of TPT has been sub-optimal globally particularly in children. A safe and effective short-course TPT regimen, 3HP (rifapentine and isoniazid given once weekly for three months), is available but there is a lack of child-friendly formulations resulting in increased pill burden and there is a need to improve acceptability and adherence among children. The introduction of a dispersible rifapentine formulation has potential to improve uptake, treatment adherence and completion.

Overall goal is to generate critical knowledge to improve delivery of TPT and, more specifically, of dispersible 3HP, in children in routine programs.

This evaluation will create an important understanding of TPT uptake and completion among children and assess the impact of the introduction of a dispersible 3HP formulation. These results will provide actionable information for improving service delivery and the scale-up of TPT in the respective countries.

ELIGIBILITY:
Clinic record review

Inclusion Criteria:

* Medical records of children <12 years who are either CLHIV or who are household contacts of people with pulmonary TB and who are initiated on TPT

Exclusion Criteria:

* Records will be excluded for children who are contacts of a drug-resistant, have presumptive TB disease or are currently on TB treatment

Qualitative study

Inclusion Criteria:

* Adult caregiver (>18 years) of a child <12 years of age who is eligible for TPT
* Healthcare worker from one of the clinics in which the study will be conducted who sees outpatient pediatric consultations including TB-exposed children
* Policy maker or program manager who manages or is involved in PMTCT, TB and/or pediatric programming

Exclusion Criteria:

* Any adult caregivers, healthcare workers, policy makers or program managers who are unable or unwilling to provide informed consent for both the interview and audio-recording.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clinic record review: Routine program data for CLHIV <12 years or children <12 years who are household contacts of people living with TB, who are initiated on TPT.
  [A household contact is defined as a person who shared the same enclosed living space with the index patient (someone with infectious TB as defined by country guidelines) for one or more nights or for frequent or extended periods during the day during the 3 months before commencement of the current treatment episode.]
  Qualitative study: Policy makers, healthcare workers and parents/caregivers will be interviewed - (>18 years)
  Clinic-level assessment: Pharmacy managers/pharmacists, procurement and supply management staff - (>18 years)
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Overarching Objective | 18 months
  The overarching goal of the evaluation is to generate critical knowledge to improve delivery of TPT and, more specifically, of dispersible 3HP, in children in routine programs.
Primary Objective 1 | 18 months
  To quantify the TPT care cascade from identification, screening, eligibility, treatment initiation to completion among children <12 years of age, stratified by regimen.

SECONDARY OUTCOMES:
Secondary Objective 1 | 18 months
  To quantify the prescription of the new dispersible 3HP vs other regimens among children <12 years.
Secondary Objective 2 | 18 months
  To explore policy makers, healthcare workers and caregivers' insights on different regimens and formulations.
Secondary Objective 3 | 18 months
  To assess provider-level barriers and facilitators to delivery of the new dispersible 3HP regimen.
Secondary Objective 4 | 18 months
  To determine the impact of the new dispersible 3HP on supply chain and changes needed to accommodate them.

OTHER OUTCOMES:
Outcome 1 | 18 months
  Any uptake of TPT defined as proportion of eligible children who are initiated on TPT, stratified by regimen
Outcome 2 | 18 months
  Proportion of children <12 years initiated on TPT who complete treatment, stratified by regimen.
Outcome 3 | 18 months
  Caregiver experience with and attitudes towards the new dispersible 3HP formulation.
Outcome 4 | 18 months
  Barriers and facilitators of the new dispersible 3HP experienced by healthcare workers and policy makers.
Outcome 5 | 18 months
  Logistics and supply chain issues related to country level procurement, forecasting and distribution to clinic level for the dispersible 3HP.

IPD SHARING:
Plan to Share IPD: Undecided
The evaluation findings will be presented at stakeholder meetings at national level and disseminated to stakeholders and participating sites in each country by means of local meetings. Results will also be written up as conference abstracts and/or journal articles and submitted for publication to an appropriate journal to maximise their dissemination, particularly to clinicians involved in TB programmes.